CLINICAL TRIAL: NCT06145425
Title: Testing an Evidence-Based Program for Physician and Nurse Burnout
Brief Title: Testing an Evidence-Based Program for Clinician Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Peter G. Peterson Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: "IRB #2022003296"
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Burnout
Keywords: Burnout; Mindfulness; Physicians; Nurses; Resident Physicians
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: 3 single groups: physicians, resident physicians and nurses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Participants will be asked to utilize the app.
  Interventions: Other: App-Delivered Mindfulness Training (MT)

INTERVENTIONS:
Other: App-Delivered Mindfulness Training (MT) — The program is delivered via a smartphone-based platform, which includes 7 mindfulness-based modules of about 15 minutes of brief didactic and experience-based mindfulness training (audio files).

SUMMARY:
The goal of this clinical trial is to pilot test an app-based mindfulness training program in reducing burnout in physicians and nurses.

DETAILED DESCRIPTION:
The main question[s] it aims to answer are:

PRIMARY AIM: Determine if the app-based training reduces the level of cynicism (i.e., one of the two main dimensions of burnout).

SECONDARY AIM: Determine if the app-based training reduces the level of emotional exhaustion (i.e. one of the two main dimensions of burnout), anxiety, worry, depression and intolerance of uncertainty. Determine if the app-based training increases self-compassion, non-reactivity and non-judging about inner experiences.

Participants will be asked to:

* Use an app-based mindfulness training program
* Complete online surveys at baseline, immediately post-intervention and 1 month after the post-intervention as follow up

ELIGIBILITY:
Inclusion Criteria:

* Being a physician, resident physician or nurse
* Able to speak English because all study activities will be conducted in English.
* 18+ years
* direct patient care

Exclusion Criteria:

* If using psychotropic medication - not on a stable dosage at least 6 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Changes in cynicism | collected at baseline, immediately post-intervention and one month later as follow up
  The dimension of cynicism in the Maslach Burnout Inventory (MBI) cynicism. The MBI is a validated 22-item self-report measure of risk of burnout. Items are rated on a 7-point Likert scale ranging from 0 (never) to 6 (every day). The investigators will use only one single-item measure of cynicism that was included from the Maslach Burnout Inventory (MBI).

SECONDARY OUTCOMES:
The dimension of emotional exhaustion in the Maslach Burnout Inventory (MBI). | collected at baseline, immediately post-intervention and one month later as follow up
  The MBI is a validated 22-item self-report measure of risk of burnout. Items are rated on a 7-point Likert scale ranging from 0 (never) to 6 (every day). The investigators will use only one single-item measure of emotional exhaustion that was included from the Maslach Burnout Inventory (MBI).
Generalized Anxiety Disorder 7-items (GAD-7). | collected at baseline, immediately post-intervention and one month later as follow up
  The GAD-7 is a validated 7-item measure of anxiety rated on a 4-point Likert scale ranging from 0 (Not at all sure) to 3 (Nearly every day).
Five Facet Mindfulness Questionnaire (FFMQ) non-reactivity scale. | collected at baseline, immediately post-intervention and one month later as follow up
  The non-reactivity scale is a validated subscale of the 39-item FFMQ which is a self-report psychological measure of mindfulness skills. This subscale contains 7 items which are presented on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never).
Five Facet Mindfulness Questionnaire (FFMQ) non-judging scale. | collected at baseline, immediately post-intervention and one month later as follow up
  The non-judging scale is a validated subscale of the 39-item FFMQ which is a self-report psychological measure of mindfulness skills. This subscale contains 8 items which are presented on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never).
Patient Health Questionnaire 2-item scale (PHQ-2). | collected at baseline, immediately post-intervention and one month later as follow up
  The PHQ-2 is a validated 2-item self-report measure of depression. Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
Penn State Worry Questionnaire (PSWQ). | collected at baseline, immediately post-intervention and one month later as follow up
  The PSWQ is a validated 16-item self-report measure of worry with items presented on a 5-point Likert scale ranging from 1 (not at all typical of me) to 5 (very typical of me).
Intolerance of Uncertainty 12-item scale (IUS-12). | collected at baseline, immediately post-intervention and one month later as follow up
  The IUS-12 is a validated 12-item self-report measure of intolerance of uncertainty. Items are rated on a 5-point Likert scale ranging from 1 (not at all characteristic of me) to 5 (entirely characteristic of me).
Self-Compassion Scale - Short Form (SCS-SF). | collected at baseline, immediately post-intervention and one month later as follow up
  The SCS-SF is a validated 12-item self-report measure of self-compassion. Items are rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always).

OTHER OUTCOMES:
Demographics. | collected at baseline
  Age, gender, employment, race, ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, MD, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antico L, Brewer J. Digital Mindfulness Training for Burnout Reduction in Physicians: Clinician-Driven Approach. JMIR Form Res. 2025 Jan 24;9:e63197. doi: 10.2196/63197. PMID 39854701